CLINICAL TRIAL: NCT00865527
Title: Randomized Comparison of Virtual Colonoscopy, Optical Colonoscopy, and Fecal Occult Blood Testing for Colorectal Cancer Screening: a Pilot Study
Brief Title: Pilot Study of Colon Cancer Screening Tests
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of ongoing funding
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, John You, Assistant Professor, McMaster University
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CTC1.0
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer; Colon Cancer; Adenomatous Polyps
Keywords: Colorectal cancer; Colon cancer; Adenomatous polyps; Screening; Fecal occult blood test; Computed tomographic colonography; Colonoscopy
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Adenomatous Polyps | interventions — Occult Blood; Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fecal Occult Blood Test (Active Comparator): fecal occult blood test
  Interventions: Other: Fecal occult blood test
- Virtual Colonoscopy (Active Comparator): virtual colonoscopy
  Interventions: Procedure: Virtual colonoscopy
- Optical Colonoscopy (Active Comparator): optical (conventional / endoscopic) colonoscopy
  Interventions: Procedure: Optical colonoscopy

INTERVENTIONS:
Other: Fecal occult blood test — FOBT
  Other Names: FOBT
  Arms: Fecal Occult Blood Test
Procedure: Virtual colonoscopy — computed tomographic colonography
  Other Names: CT colonography; computed tomographic colonography
  Arms: Virtual Colonoscopy
Procedure: Optical colonoscopy — optical (conventional / endoscopic) colonoscopy
  Other Names: Colonoscopy
  Arms: Optical Colonoscopy

SUMMARY:
Colon cancer is the second leading cause of cancer death in North America. These deaths are preventable with proper screening. Fecal occult blood testing, virtual colonoscopy, and standard (optical) colonoscopy are all options for colon cancer screening, but it is not known which is the best at preventing death from colon cancer. A large study comparing these three tests is desperately needed. In this pilot study, the investigators want to find out what percentage of patients will show up for their screening test once enrolled. This will provide crucial information for the successful execution of the larger study.

ELIGIBILITY:
Inclusion Criteria:

* All individuals age 50 to 70 years

Exclusion Criteria:

* Unable to give informed consent
* History of colorectal cancer
* History of adenomatous polyp
* History of inflammatory bowel disease
* Prior participation in FOBT screening
* Prior refusal to participate in FOBT screening
* Flexible sigmoidoscopy within the previous 3 years
* Virtual colonoscopy within the previous 3 years
* Optical colonoscopy within the previous 3 years
* Severe of terminal illness that would preclude benefit from colon cancer screening

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Proportion of enrolled patients who attend for their assigned screening test | Immediate

SECONDARY OUTCOMES:
Proportion of non-responders to mailed invitations, who respond to telephone or mail reminders. | Immediate
Proportion of patients requiring polypectomy after virtual colonoscopy who receive same or next day optical colonoscopy for polypectomy | 6 months
Proportion of subjects who cross over to another arm of the study | 6 months
Proportion of patients found to have an advanced adenoma | 6 months
Proportion of patients found to have invasive colorectal carcinoma | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John J You, MD MSc FRCPC, Principal Investigator — McMaster University
Locations (1):
- Hamilton Health Sciences, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] You JJ, Liu Y, Kirby J, Vora P, Moayyedi P. Virtual colonoscopy, optical colonoscopy, or fecal occult blood testing for colorectal cancer screening: results of a pilot randomized controlled trial. Trials. 2015 Jul 9;16:296. doi: 10.1186/s13063-015-0826-7. PMID 26156248
- [Derived] Wong AD, Kirby J, Guyatt GH, Moayyedi P, Vora P, You JJ. Randomized controlled trial comparing telephone and mail follow-up for recruitment of participants into a clinical trial of colorectal cancer screening. Trials. 2013 Feb 11;14:40. doi: 10.1186/1745-6215-14-40. PMID 23399518